CLINICAL TRIAL: NCT04719351
Title: Diary of a Pandemic: The Use of a Mobile Application to Reduce Work-related Stress Symptoms Among Healthcare Workers
Brief Title: The Use of a Mobile Application to Reduce Work-related Stress Symptoms Among Healthcare Workers
Acronym: DIARY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Aleksandra Sjöström-Bujacz, Project Leader, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 4-2092/2020; 2020-05800 (Other: The Swedish Research Council (VR))
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Burnout, Professional; Stress, Psychological
Keywords: mobile application; healthcare workers; work stress
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Occupational Stress

STUDY DESIGN:
Intervention Model Description: The factorial experimental trial will randomize participants to one of 32 experimental conditions which consist of any combination of the five components: 1) questions about positive emotions (yes/no), 2) questions about work environment (yes/no), 3) questions about controllability (yes/no), 4) questions with open answers (yes/no), and 5) behavioral prompts (yes/no). The purpose of this factorial experiment is to estimate the main effects of the five intervention components and interactions between the components.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Condition 1: Positive: no; Workload: no; Controllability: no; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 2: Positive: yes; Workload: no; Controllability: no; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 3: Positive: no; Workload: yes; Controllability: no; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 4: Positive: yes; Workload: yes; Controllability: no; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 5: Positive: no; Workload: no; Controllability: yes; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 6: Positive: yes; Workload: no; Controllability: yes; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 7: Positive: no; Workload: yes; Controllability: yes; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 8: Positive: yes; Workload: yes; Controllability: yes; Open: no; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 9: Positive: no; Workload: no; Controllability: no; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 10: Positive: yes; Workload: no; Controllability: no; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 11: Positive: no; Workload: yes; Controllability: no; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 12: Positive: yes; Workload: yes; Controllability: no; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 13: Positive: no; Workload: no; Controllability: yes; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 14: Positive: yes; Workload: no; Controllability: yes; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 15: Positive: no; Workload: yes; Controllability: yes; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 16: Positive: yes; Workload: yes; Controllability: yes; Open: yes; Prompt: no; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: not included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 17: Positive: no; Workload: no; Controllability: no; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 18: Positive: yes; Workload: no; Controllability: no; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 19: Positive: no; Workload: yes; Controllability: no; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 20: Positive: yes; Workload: yes; Controllability: no; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 21: Positive: no; Workload: no; Controllability: yes; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 22: Positive: yes; Workload: no; Controllability: yes; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 23: Positive: no; Workload: yes; Controllability: yes; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 24: Positive: yes; Workload: yes; Controllability: yes; Open: no; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: not included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 25: Positive: no; Workload: no; Controllability: no; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 26: Positive: yes; Workload: no; Controllability: no; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 27: Positive: no; Workload: yes; Controllability: no; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 28: Positive: yes; Workload: yes; Controllability: no; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: not included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 29: Positive: no; Workload: no; Controllability: yes; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 30: Positive: yes; Workload: no; Controllability: yes; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: not included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 31: Positive: no; Workload: yes; Controllability: yes; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: not included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application
- Condition 32: Positive: yes; Workload: yes; Controllability: yes; Open: yes; Prompt: yes; (Experimental): Component list:
  1. Questions about positive emotions: included;
  2. Questions about workload/work environment: included;
  3. Questions about controllability: included;
  4. Questions with open answers: included;
  5. Behavioral prompts: included;
  Interventions: Behavioral: The DIARY mobile application

INTERVENTIONS:
Behavioral: The DIARY mobile application — The mobile application has two main functionalities. First, it will remind the user to report in regular time periods on their mental health status (e.g., sleep disturbances, stress). The assessment is done daily for four weeks. Second, some completed assessments will be combined with a behavioral prompt i.e. short message encouraging the user to engage in one of the strategies that can help coping with stress at work, e.g. remember to take short breaks, exercise in daylight, summarize a day with a colleague after a finished shift.

SUMMARY:
The current pandemic highlighted an urgent need for early interventions to mitigate the psychological effects of extreme work demands that healthcare workers currently experience. This project aims at developing a data driven monitoring system to efficiently track work-related stress reactions over time. The system will also include a self-awareness intervention grounded on evidence-based strategies to improve workers' recovery. The solution will be delivered through a mobile application for a rapid implementation among healthcare workers and related professions. The mobile application will be developed through an initial analysis of pilot data, a factorial experiment and a user-experience analysis. Qualitative user experience data will also be used to validate the functionality of the monitoring system. The solution developed in this project will be easily scalable to related occupations, for example workers at elderly homes and social workers. After the pandemic, it can also be used as a preventive intervention for workers who are at risk of burnout and as a support for patients returning to work after treatment for common mental disorders.

DETAILED DESCRIPTION:
Symptoms indicating possibly pathological stress reactions among healthcare workers are more prevalent during the current pandemic than they were before. Possible reasons for that include higher levels of known risk factors such as cognitive, emotional, and physical demands at work; new stressors such as risk for moral injury and worry about personal safety; and diminished protective mechanisms, which include recovery opportunities and psychological detachment. Thus, frontline healthcare workers should be given priority in access to psychological support.

Despite the urgent need for it, a rapid implementation of psychological support for healthcare workers has proved to be challenging during previous crises and the current pandemic. Guidelines published thus far underline the necessity of close real-time monitoring in order to early identify at risk populations and individuals, who should be referred to seek professional support. However, appropriate tools for efficient real-time monitoring of stress responses and early screening for possibly pathological reactions among healthcare workers are currently lacking. Available tools focus either on tracking of stress indicators e.g. sleep disturbances, or on teaching strategies to better cope with stress e.g. mindfulness.

In this study, the investigators will test whether a separate use or a combination of these different functions may be the most efficient in managing work-related stress symptoms among healthcare workers. The study has a factorial design in order to closely investigate the functionalities focused on real-time monitoring of emotional responses and the functionalities based on evidence-based strategies to improve workers' recovery, as well as the possible interactions among them.

ELIGIBILITY:
Inclusion Criteria:

* adult participants
* working (active employment)

Exclusion Criteria:

- no active employment e.g. sick leave, maternity leave during the entire period of an intervention (four weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Burnout symptoms immediate effect | Immediately post-intervention
  Burnout is measured using Oldenburg Burnout Inventory (Olbi), an instrument designed to measure exhaustion and disengagement: (Demerouti, E, Bakker, A.B, Vardakou, I, & Kantas, A. [2003]. The convergent validity of two burnout instruments : a multitrait-multimethod analysis. European Journal of Psychological Assessment : Official Organ of the European Association of Psychological Assessment, 19(1), 12-23. https://doi.org/10.1027//1015-5759.19.1.12)
  The full Olbi scale consists of twelve items, and this study uses a subset of seven items. The study uses a Swedish version: Gustavsson, J. P., Hallsten, L., & Rudman, A. (2010). Early career burnout among nurses: modelling a hypothesized process using an item response approach. International Journal of Nursing Studies, 47(7), 864-875.
  The items are scored on a 4-point Likert scale (1 = Not at all, 4 = Exactly).
Burnout symptoms delayed effect | A month after completed intervention
  Burnout is measured using Oldenburg Burnout Inventory (Olbi), an instrument designed to measure exhaustion and disengagement: (Demerouti, E, Bakker, A.B, Vardakou, I, & Kantas, A. [2003]. The convergent validity of two burnout instruments : a multitrait-multimethod analysis. European Journal of Psychological Assessment : Official Organ of the European Association of Psychological Assessment, 19(1), 12-23. https://doi.org/10.1027//1015-5759.19.1.12)
  The full Olbi scale consists of twelve items, and this study uses a subset of seven items. The study uses a Swedish version: Gustavsson, J. P., Hallsten, L., & Rudman, A. (2010). Early career burnout among nurses: modelling a hypothesized process using an item response approach. International Journal of Nursing Studies, 47(7), 864-875.
  The items are scored on a 4-point Likert scale (1 = Not at all, 4 = Exactly).
Emotional exhaustion immediate effect | Immediately post-intervention
  Emotional exhaustion is measured using Shirom-Melamed Burnout questionnaire (SMBQ), a 22-item instrument designed to assess burnout: Shirom, A., & Melamed, S. (2006). A comparison of the construct validity of two burnout measures in two groups of professionals. International journal of stress management, 13(2), 176.
  This study uses the SMBQ-6, a subset of six items, specifically measuring emotional exhaustion. A Swedish version is used for this study: Lundgren-Nilsson, Å., Jonsdottir, I. H., Pallant, J., & Ahlborg, G. (2012). Internal construct validity of the Shirom-Melamed Burnout questionnaire (SMBQ). BMC public health, 12(1), 1.
  Items are scored on a 7-point Likert scale (1 = Very rarely, 7 = Very frequently).
Emotional exhaustion delayed effect | A month after completed intervention
  Emotional exhaustion is measured using Shirom-Melamed Burnout questionnaire (SMBQ), a 22-item instrument designed to assess burnout: Shirom, A., & Melamed, S. (2006). A comparison of the construct validity of two burnout measures in two groups of professionals. International journal of stress management, 13(2), 176.
  This study uses the SMBQ-6, a subset of six items, specifically measuring emotional exhaustion. A Swedish version is used for this study: Lundgren-Nilsson, Å., Jonsdottir, I. H., Pallant, J., & Ahlborg, G. (2012). Internal construct validity of the Shirom-Melamed Burnout questionnaire (SMBQ). BMC public health, 12(1), 1.
  Items are scored on a 7-point Likert scale (1 = Very rarely, 7 = Very frequently).
Stress symptoms immediate effect | Immediately post-intervention
  Stress is measured using the Perceived Stress Scale (PSS), designed to measure "the degree to which situations in one´s life are appraised as stressful" (Cohen, S., Kamarck, T., & Mermelstein, R. [1983]. A global measure of perceived stress. Journal of health and social behavior, 385-396).
  The original scale contains 14 items, and this study uses the PSS-10 version which contains 10 items. A Swedish translation of the scale is used: Nordin, M., & Nordin, S. (2013). Psychometric evaluation and normative data of the Swedish version of the 10-item perceived stress scale. Scandinavian journal of psychology, 54(6), 502-507.
  The items are scored on a 5-point Likert scale (1 = Never, 5 = Very often).
Stress symptoms delayed effect | A month after completed intervention
  Stress is measured using the Perceived Stress Scale (PSS), designed to measure "the degree to which situations in one´s life are appraised as stressful" (Cohen, S., Kamarck, T., & Mermelstein, R. [1983]. A global measure of perceived stress. Journal of health and social behavior, 385-396).
  The original scale contains 14 items, and this study uses the PSS-10 version which contains 10 items. A Swedish translation of the scale is used: Nordin, M., & Nordin, S. (2013). Psychometric evaluation and normative data of the Swedish version of the 10-item perceived stress scale. Scandinavian journal of psychology, 54(6), 502-507.
  The items are scored on a 5-point Likert scale (1 = Never, 5 = Very often).

SECONDARY OUTCOMES:
Anxiety symptoms immediate effect | Immediately post-intervention
  Anxiety is measured using the GAD-7 scale, a 7-item questionnaire designed to assess generalized anxiety disorder (Spitzer, R. L., Kroenke, K., Williams, J. B., & Löwe, B. [2006]. A brief measure for assessing generalized anxiety disorder: the GAD-7. Archives of internal medicine, 166(10), 1092-1097). A Swedish version of the scale will be used.
  The items are scored on a 4-point Likert scale (1 = Not at all, 4 = Almost every day).
Anxiety symptoms delayed effect | A month after completed intervention
  Anxiety is measured using the GAD-7 scale, a 7-item questionnaire designed to assess generalized anxiety disorder (Spitzer, R. L., Kroenke, K., Williams, J. B., & Löwe, B. [2006]. A brief measure for assessing generalized anxiety disorder: the GAD-7. Archives of internal medicine, 166(10), 1092-1097). A Swedish version of the scale will be used.
  The items are scored on a 4-point Likert scale (1 = Not at all, 4 = Almost every day).
Depressive symptoms immediate effect | Immediately post-intervention
  Depressive symptoms are measured using the Patient Health Questionnaire-2 (PHQ-2), a 2-item screening tool for assessing depression (Kroenke, K., Spitzer, R. L., & Williams, J. B. [2003]. The Patient Health Questionnaire-2: validity of a two-item depression screener. Medical care, 1284-1292). A Swedish translation is used.
  The items are scored on a 4-point Likert scale (1 = Not at all, 4 = Almost every day)
Depressive symptoms delayed effect | A month after completed intervention
  Depressive symptoms are measured using the Patient Health Questionnaire-2 (PHQ-2), a 2-item screening tool for assessing depression (Kroenke, K., Spitzer, R. L., & Williams, J. B. [2003]. The Patient Health Questionnaire-2: validity of a two-item depression screener. Medical care, 1284-1292). A Swedish translation is used.
  The items are scored on a 4-point Likert scale (1 = Not at all, 4 = Almost every day)
Post-traumatic stress immediate effect | Immediately post-intervention
  PTSD is measured using the Posttraumatic Stress Disorder checklist (PCL-5), a widely used self-report measure of PTSD using criteria from the DSM-5 (Bovin, M. J., Marx, B. P., Weathers, F. W., Gallagher, M. W., Rodriguez, P., Schnurr, P. P., & Keane, T. M. [2015]. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in Veterans. Psychological Assessment, 28, 1379-1391. doi:10.1037/pas0000254).
  The entire scale contains 20 items, and a subset of three items is used for this study. A Swedish version is used.
  Items are scored on a 5-item Likert scale (1 = A lot, 5 = Not at all).
Post-traumatic stress delayed effect | A month after completed intervention
  PTSD is measured using the Posttraumatic Stress Disorder checklist (PCL-5), a widely used self-report measure of PTSD using criteria from the DSM-5 (Bovin, M. J., Marx, B. P., Weathers, F. W., Gallagher, M. W., Rodriguez, P., Schnurr, P. P., & Keane, T. M. [2015]. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in Veterans. Psychological Assessment, 28, 1379-1391. doi:10.1037/pas0000254).
  The entire scale contains 20 items, and a subset of three items is used for this study. A Swedish version is used.
  Items are scored on a 5-item Likert scale (1 = A lot, 5 = Not at all).
Emotional awareness immediate effect | Immediately post-intervention
  Awareness of emotions is measured using Mindful Attention Awareness Scale (MAAS) (Brown, K. W., & Ryan, R. M. [2009]. The Mindfulness Attention Awareness Scale (MAAS). Acceptance and Commitment Therapy. Measures Package, 82). This study uses a subset of six questions, focusing on emotional awareness. A Swedish version is used in this study. Items are rated on a 6-point Likert scale (1 = Very frequently, 6 = Very rarely).
Emotional awareness delayed effect | A month after completed intervention
  Awareness of emotions is measured using Mindful Attention Awareness Scale (MAAS) (Brown, K. W., & Ryan, R. M. [2009]. The Mindfulness Attention Awareness Scale (MAAS). Acceptance and Commitment Therapy. Measures Package, 82). This study uses a subset of six questions, focusing on emotional awareness. A Swedish version is used in this study. Items are rated on a 6-point Likert scale (1 = Very frequently, 6 = Very rarely).
Controllability immediate effect | Immediately post-intervention
  Controllability is measured using the "control" subscale from the Recovery Experience Questionnaire (REQ) (Sonnentag, S., & Fritz, C. [2007]. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. Journal of occupational health psychology, 12(3), 204). This subscale includes 4 items that are scored on a 5-point Likert scale (1 = Not at all, 5 = Very much). A Swedish version is used.
  To measure controllability in the work context, the study also uses the Task Crafting subscale from the Job Crafting Questionnaire (Slemp, G. R., & Vella-Brodrick, D. A. [2013]. The Job Crafting Questionnaire: A new scale to measure the extent to which employees engage in job crafting. International Journal of wellbeing, 3(2)). A Swedish version is used. This subscale includes 7 items scored on a 5-point Likert scale (1 = Hardly ever, 5 = Very often).
Controllability delayed effect | A month after completed intervention
  Controllability is measured using the "control" subscale from the Recovery Experience Questionnaire (REQ) (Sonnentag, S., & Fritz, C. [2007]. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. Journal of occupational health psychology, 12(3), 204). This subscale includes 4 items that are scored on a 5-point Likert scale (1 = Not at all, 5 = Very much). A Swedish version is used.
  To measure controllability in the work context, the study also uses the Task Crafting subscale from the Job Crafting Questionnaire (Slemp, G. R., & Vella-Brodrick, D. A. [2013]. The Job Crafting Questionnaire: A new scale to measure the extent to which employees engage in job crafting. International Journal of wellbeing, 3(2)). A Swedish version is used. This subscale includes 7 items scored on a 5-point Likert scale (1 = Hardly ever, 5 = Very often).
Recovery experience immediate effect | Immediately post-intervention
  Questions regarding the degree to which participants engage in behavioral recovery strategies, for instance spending time on a hobby or letting go of work-related thoughts. This is measured using the Recovery Experience Questionnaire (REQ) (Sonnentag, S., & Fritz, C. [2007]. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. Journal of occupational health psychology, 12(3), 204). The study uses two subscales - psychological detachment and relaxation, resulting in 8 items. Items are scored on a 5-point Likert scale (1 = Not at all, 5 = Very much). A Swedish version is used.
Recovery experience delayed effect | A month after completed intervention
  Questions regarding the degree to which participants engage in behavioral recovery strategies, for instance spending time on a hobby or letting go of work-related thoughts. This is measured using the Recovery Experience Questionnaire (REQ) (Sonnentag, S., & Fritz, C. [2007]. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. Journal of occupational health psychology, 12(3), 204). The study uses two subscales - psychological detachment and relaxation, resulting in 8 items. Items are scored on a 5-point Likert scale (1 = Not at all, 5 = Very much). A Swedish version is used.
Social support immediate effect | Immediately post-intervention
  Questions regarding the degree to which participants engage with their social context for emotional support. We use the Relation Crafting subscale from the Job Crafting Questionnaire: (Slemp, G. R., & Vella-Brodrick, D. A. (2013). The Job Crafting Questionnaire: A new scale to measure the extent to which employees engage in job crafting. International Journal of wellbeing, 3(2)). The subscale includes 7 items scored on a 5-point Likert scale (1 = Hardly ever, 5 = Very often).
Social support delayed effect | A month after completed intervention
  Questions regarding the degree to which participants engage with their social context for emotional support. We use the Relation Crafting subscale from the Job Crafting Questionnaire: (Slemp, G. R., & Vella-Brodrick, D. A. (2013). The Job Crafting Questionnaire: A new scale to measure the extent to which employees engage in job crafting. International Journal of wellbeing, 3(2)). The subscale includes 7 items scored on a 5-point Likert scale (1 = Hardly ever, 5 = Very often).

OTHER OUTCOMES:
Dropout rate | Immediately post-intervention
  Investigates the dropout rate during the four weeks of the intervention.
Protocol adherence | Immediately post-intervention
  Investigates how often (i.e. how many days) participants engage with the intervention.
Participant engagement | Immediately post-intervention
  Investigates to what extent participants engage with the intervention, as measured with the meta-data available through the mobile application e.g. time spent engaging with the content of the mobile application.
Usability: User experience, relevance, and content appreciation | Immediately post-intervention
  Investigates basic usability questions in a post-intervention survey. Includes questions about the experience users had of using the mobile application, if they found the intervention relevant, and if they found the content useful.
  Survey questions focus on specific aspects of the mobile application used in this study. The survey includes 10 items scored on a 4-point Likert scale. High scores refer to higher usability, relevance and content appreciation.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Sjostrom-Bujacz, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Aleksandra Sjostrom-Bujacz, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
An anonymized subset of the data relevant for a particular publication (including metadata and code for the analyses conducted) will be registered on the OSF repository and provided with the DOI number. Neither qualitative data (i.e. answers to open questions) nor any personal data (i.e. gender, age, occupation) will be shared to ensure complete anonymity of the study participants. Data regarding each publication will become available already at the pre-print stage of each publication (i.e. manuscript submitted for publication), under the CC-BY license. Data will be stored in .csv format and will include raw data as well as data analysis files (analysis code). The data publication may be postponed and restricted in case a patent application will be submitted for a review.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will become available upon each scientific publication, at the preprint stage. Complete anonymized dataset will be shared no later than four years after initial data collection took place.
Access Criteria: Anyone can view.
URL: https://osf.io/uz3b7/?view_only=ba37189d0b594529b159ba27564dfb81

REFERENCES:
- Available data/document: Individual Participant Data Set — https://osf.io/uz3b7/?view_only=ba37189d0b594529b159ba27564dfb81